CLINICAL TRIAL: NCT06924437
Title: Evaluation of the Uterine Cavity After Operative Hysteroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Allam Mohamed, Resident, Sohag University
Other Study IDs: Soh-Med--25-3-05MS
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Uterine Abnominalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will focus on evaluation of the uterine cavity after operative hysteroscopy using three-dimentional tranvaginal ultrasonography and office hysteroscopy to detect and residual or recurrent abnormalities or intrauterine adhesions to optimize the results of operatve hysteroscopy in different uterine pathologies such as uterine polyps, fibroids, adhesions in addition to mullerian anomalies especially septate uteri.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in reproductive age group
2. Patients already selected for operative hysteroscopy
3. Patients accepted to share in the study
4. Patients accepted to come for follow up ( within 3 months after the initial operative procedure, at least after 4 weeks

Exclusion Criteria:

1. Patients outside the age of reproduction
2. Patients with negative findings at operative hysteroscopy
3. Patients refused to share in the study
4. Patients not available for follow up
5. Infection
6. pregnancy or design of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological females
Study Population: It will be held in the department of Obstetrics and Gynecology during the period from February 2025 to February 2026. The study will include all recruited patients who will be selected for operative hysteroscopy during that period.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
1- accuracy | one year
  Comparing thee- dimentional ultrasonography and office hysteroscopy for uterine cavity evaluation after operatve hysteroscopy as regards accuracy, pain score, and cost-effectiveness of each method.